CLINICAL TRIAL: NCT01506245
Title: Exercise Training and Family-based Behavioural Treatment in Pre-pubertal Obese Children and Their Mother
Brief Title: Exercise and Behavioral Therapy in Obese Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University Hospital, Geneva (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Principal Investigator, Nathalie Farpour-Lambert, Head of the Obesity Care Program, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNF 3200B0-120437
Record Dates: First submitted 2011-12-31; First posted 2012-01-09 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2012-01

CONDITIONS: Childhood Obesity
Keywords: Obesity; Children; Behavior; Family; Exercise
MeSH Terms: conditions — Pediatric Obesity; Obesity; Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention)
- Family-based behavioral therapy (Experimental): Family-based behavioural therapy either in group or in individual setting. Parents can choose between the 2 types of therapy.
  Interventions: Behavioral: Family-based behavioral therapy

INTERVENTIONS:
Behavioral: Family-based behavioral therapy — The intervention consist of a 6-month family-based behavioural therapy either in group (1 session/week, with a dietician and a psychologist) or in individual setting (with a paediatrician or a dietician in alternance 1x/month). Both therapies include exercise training twice per week (60 minutes each). Parents, or at at least the mother, must participate to the behavioral treatment.
  Arms: Family-based behavioral therapy

SUMMARY:
The aim of this study is to compare the effects of exercise training and family-based behavioral treatment, either in individual or in group setting, in pre-pubertal children and their mother.

DETAILED DESCRIPTION:
Introduction: The prevalence of childhood obesity is increasing rapidly in developing countries. The aim of this study is to determine the effects of exercise training and family-based behavioral treatment (FBBT), either in individual or in group setting,in pre-pubertal children and their mother.

Methods: This is a 6-month randomized controlled trial (RCT) including 75 pre-pubertal obese children (age 8-11 years) randomly assigned to an Intervention (I, n=50) or a Control group (C, n=25). The intervention consists of a family-based behavioural therapy in group (1 session/week with a dietician and a psychologist) or in individual setting (paediatrician or dietician 1x/month). The intervention includes exercise training sessions twice a week (60 minutes each).

Measures include: body mass index (BMI), waist and hip circumferences; whole body and abdominal fat mass by DXA; resting and ambulatory blood pressure; arterial intima-media thickness and vascular reactivity (flow-mediated dilation)using high resolution ultrasound; arterial stiffness by tonometry of applanation; cardiorespiratory fitness by a treadmill test; physical activity; fasting lipids, glucose, insulin, and C-reactive protein levels; health-related quality of life and psychological health using standardized questionnaires and a semi-structured interview. Measures are completed in children and their mother at baseline and 6 months post-randomization.

ELIGIBILITY:
Inclusion Criteria:

* Childhood obesity (>97 percentile WHO references)

Exclusion Criteria:

* being involved in any weight control, physical activity, behavior therapy, or gastric surgery program;
* familial history of dyslipidemia or essential hypertension;
* medications or hormones, which may influence cardiovascular function, body composition, lipid or glucose metabolism in the preceding 6 months;
* orthopaedic affection limiting physical activity;
* genetic disorder or another chronic disease;

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2011-01; Primary Completion 2012-06 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Body Mass Index at 6 months | 6 months
  Body Mass Index (weight/height 2) expressed in Standard Deviation Score

SECONDARY OUTCOMES:
Change from baseline in total body and abdominal fat at 6 months | 6 months
  Body fat mass and percentage assessed using DXA
Change from baseline in waist circumference at 6 months | 6 months
Change from baseline in blood pressure at 6 months | 6 months
  Resting and ambulatory (24 hours) systolic and diastolic blood pressure
Change from baseline in arterial intima-media thickness at 6 months | 6 months
  Measure of the arterial intima-media thickness using high-resolution ultrasound
Change from baseline in arterial flow-mediated dilation at 6 months | 6 months
  Measure of the flow-mediated dilation of the brachial artery using high-resolution ultrasound
Change from baseline in arterial stiffness at 6 months | 6 months
  Measure of mechanical indices using tonometry of applanation
Change from baseline in cardiorespiratory fitness at 6 months | 6 months
Change from baseline in physical activity at 6 months | 6 months
  Physical activity pattern using accelerometer
Change from baseline in biological markers at 6 months | 6 months
  Fasting glucose, insulin, total-, LDL-, HDL-cholesterol, high-sensitive C-reactive protein.
Change from baseline in quality of life at 6 months | 6 months
  Quality of life assessed using the Kidsscreen 52 questionnaire
Change from baseline in child's behavior at 6 months | 6 months
  Child Behavior Checklist filled by parents
Change from baseline in parental psychological health at 6 months | 6 months
  Global Health Questionnaire filled by parents

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Farpour-Lambert, MD, Principal Investigator — University of Geneva
Locations (1):
- University Hospital of Geneva, Geneva, Canton of Geneva, Switzerland